CLINICAL TRIAL: NCT02848417
Title: Testing the Model: A Phase I/II Randomized Double Blind Placebo Control Trial of Targeted Therapeutics: Liposomal Glutathione and Curcumin
Brief Title: Glutathione vs. Curcumin Clinical Trial
Acronym: Glutathione
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Florida Veterans Affairs Foundation for Research and Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nancy Klimas, M.D, South Florida Veterans Affairs Foundation for Research and Education
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4987
Record Dates: First submitted 2016-07-06; First posted 2016-07-28 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Gulf War Syndrome
MeSH Terms: conditions — Persian Gulf Syndrome | interventions — Curcumin; Glutathione

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Curcumin (Experimental): 12 weeks 400mg orally twice a day
  Interventions: Drug: Curcumin
- Liposomal Glutathione (Experimental): 12 weeks 630mg orally twice a day
  Interventions: Drug: Glutathione
- Placebo Liquid or Capsules (Experimental): Placebo liquid for Glutathione 120 ml per/ bottle 420 mg/5 ml
  Placebo capsules for Curcumin 60 capsules per bottle 400 mg /cap
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Curcumin — Perform a randomized phase I/II study comparing curcumin (increased bioavailable form, body cell mass-85, 400 mg twice a day) to glutathione (liposomal bioavailable form 630 mg bid), with a 3 month intervention and assessment of safety, efficacy and biomarker response to therapy.
  Arms: Curcumin
Drug: Glutathione — Perform dynamic modeling studies before and after 3 months of therapy, repeating the method used previously in order to compare the response to exercise across groups and better quantify the degree of recovery in treated subjects using an exercise challenge and 9 point in time blood and saliva collections over 24 hours with genomic, cytokine, neuropeptide and cell population studies.
  Arms: Liposomal Glutathione
Other: Placebo — Placebo liquid 120 ml per/ bottle
  Placebo capsules 60 capsules per bottle 400 mg /cap
  With the addition of a Partner PI, redox/methylation expert Dr. Richard Deth, perform studies of antioxidant and methylation-related metabolic status prior to, during and after acute exercise in GWI subjects before and after interventions.
  Arms: Placebo Liquid or Capsules

SUMMARY:
The investigator proposes to perform a phase I/II study comparing two nutraceuticals and placebo that target mediators identified in the investigator's prior dynamic modeling study of Gulf War Illness (GWI). The investigator will repeat the dynamic modeling before treatment and on therapy to assess the modeling and the impact of the interventions on the homeostatic networks that have identified, with an added focus on the glutathione/redox system.

DETAILED DESCRIPTION:
In the Investigator's prior study "Dynamic Modeling in GWI", the investigator used an exercise stress model (rest, peak oxygen consumption oxygen uptake, and 7 follow-up sampling points) to measure the mediators of relapse in the context of their interactive homeostatic networks. The investigator surveyed the response of genes and blood-borne biomarkers in order to interrogate and map regulation of neuro-endocrine-autonomic-immune function in these subjects as compared to GW era sedentary healthy controls. The investigator's research team applied an integrative systems-based approach rooted in computational biology connecting gene expression and biomarkers to pathways and to symptoms in order to identify potential therapeutic targets as well as optimal strategies for manipulation of these targets. Using this data the investigator's research team has developed a virtual model of the illness, which has been used to identify potential therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with Gulf War Illness
* 35 to 70 years old
* Good health by medical history prior to 1990
* Currently have no exclusionary diagnoses that could reasonably explain the symptoms of their fatiguing illness and their severity

Exclusion Criteria:

* Major depression with psychotic or melancholic features
* Schizophrenia
* Bipolar disorder
* Delusional disorders
* Dementias of any type
* History or current alcohol abuse
* History or current drug abuse
* Current tobacco use
* Organ failure
* Defined rheumatologic
* Inflammatory disorders
* HIV
* Hepatitis B and C
* Primary sleep disorders
* Steroids
* Immunosuppressives

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2016-04; Primary Completion 2019-08 (Actual); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Biomarker response to therapy using a VO2 exercise test | 12 weeks
  Goal is that both will prove safe for use in GWI patients
Biomarker response to therapy using cytokine panel | 12 weeks
  Goal is that both will prove safe for use in GWI patients

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Balbin, Study Director — Nova University
Locations (1):
- Miami VA Center, Miami, Florida, United States